CLINICAL TRIAL: NCT00975897
Title: FOCUS 3 - A Study to Determine the Feasibility of Molecular Selection of Therapy Using KRAS, BRAF and Topo-1 in Patients With Metastatic or Locally Advanced Colorectal Cancer
Brief Title: Study of Tumor Tissue Testing in Selecting Treatment for Patients With Metastatic or Locally Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000648235; UKM-MRC-FOCUS3-CR12; EUDRACT-2008-008323-15; ISRCTN83171665; EU-20960
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2011-08

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; recurrent colon cancer; stage III colon cancer; stage IV colon cancer; adenocarcinoma of the rectum; recurrent rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Cetuximab; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin; Cytogenetic Analysis; In Situ Hybridization, Fluorescence; Gene Expression Profiling; Immunohistochemistry; Mental Status and Dementia Tests

INTERVENTIONS:
Biological: bevacizumab
Biological: cetuximab
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Drug: oxaliplatin
Genetic: RNA analysis
Genetic: cytogenetic analysis
Genetic: fluorescence in situ hybridization
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: protein expression analysis
Other: diagnostic laboratory biomarker analysis
Other: immunohistochemistry staining method
Other: questionnaire administration
Procedure: cognitive assessment

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors select the best treatment for patients and predict their response to treatment.

PURPOSE: This randomized phase II/III trial is studying how well tumor tissue testing works in selecting treatment for patients with metastatic or locally advanced colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary - Feasibility Study

* To determine the proportion of consenting patients that can provide a formalin-fixed paraffin-embedded block containing tumor.
* To determine the feasibility of topoisomerase-1 (topo-1) IHC and K-ras, BRAF mutational status determination being completed with 10 working days of initial consent.
* To determine reproducibility of results between reference laboratories.
* To determine the real costs of molecular testing.
* To determine the patients' ability to comprehend the study and their attitude during the waiting period for testing.
* To assess patients' ability to fully comprehend the trial as explained to them.

Secondary - Feasibility Study

* To further identify the EGFR-responsive subset within the K-ras wildtype population.

Primary - Definitive Study

* Compare the clinical outcomes of patients with metastatic or locally advanced colorectal cancer and low topo-1-expressing tumors treated with fluorouracil alone versus irinotecan hydrochloride, fluorouracil, and leucovorin calcium (IrMdG).
* Compare the progression-free survival of patients with high topo-1-expressing tumors treated with oxaliplatin and IrMdG versus IrMdG alone.
* Compare the response rate in patients with K-ras wildtype tumor treated with cetuximab and IrMdG versus IrMdG alone.
* Compare the response rate in patients with K-ras mutant tumors who are unlikely to respond to EGFR inhibition treated with bevacizumab and IrMdG versus IrMdG alone.

OUTLINE: This is a multicenter, 2-part study.

* Part I (feasibility study): Once consent for tissue block release has been obtained and patient is registered, the block is requested from the Pathology Department. This begins the 10 working-day time line. Treatment commences once the results of the testing are known. The following evaluations are performed during this period:

  * The frequency of EGFR gene amplification on FISH, PI3K gene mutation, PTEN loss by IHC, estimation of mRNA for EGFR ligands (amphiregulin and epiregulin), and other protein assessments.
  * An evaluation of the impact on the use or further investigation of these markers in the main study.
  * Patients consenting to trial entry and (if agreeable to data collection) patients refusing trial entry complete a questionnaire assessing patients' ability to fully comprehend the trial as explained to them.
  * Patients are interviewed before allocation of treatment about their attitudes about the waiting period necessary for tumor testing.
* Part II (definitive study): Patients are stratified according to availability of both lab tests (K-ras mutation [yes vs no], BRAF mutation [yes vs no], and topoisomerase-1 [topo-1] expression [low vs high]). Patients are assigned to 1 of 4 treatment groups based on their biomarker test results.

  * Group 1 (low topo-1 and both K-ras and BRAF wildtype): Patients are randomized to 1 of 3 treatment arms.

    * Arm I (regimen A [IrMdG]): Patients receive irinotecan hydrochloride IV over 30 minutes, leucovorin calcium IV over 2 hours, and fluorouracil IV bolus followed by infusion over 46 hours on day 1. Treatment repeats every 2 weeks for at least 6 months in the absence of disease progression or unacceptable toxicity.
    * Arm II (regimen B [MdG]): Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV bolus followed by infusion over 46 hours on day 1. Treatment repeats every 2 weeks for at least 6 months in the absence of disease progression or unacceptable toxicity.
    * Arm III (regimen D [IrMdG and cetuximab]): Patients receive cetuximab IV over 1-2 hours, irinotecan hydrochloride IV over 30 minutes, leucovorin calcium IV over 2 hours, and fluorouracil IV bolus followed by infusion over 46 hours on day 1. Treatment repeats every 2 weeks for at least 6 months in the absence of disease progression or unacceptable toxicity.
  * Group 2 (low topo-1 and either K-ras or BRAF mutation): Patients are randomized to 1 of 3 treatment arms.

    * Arm I (regimen A [IrMdG]): Patients receive irinotecan hydrochloride, leucovorin calcium, and fluorouracil as in group 1, arm I.
    * Arm II (regimen B [MdG]): Patients receive leucovorin calcium and fluorouracil as in group 1, arm II.
    * Arm III (regimen E [IrMdG and bevacizumab]): Patients receive bevacizumab IV over 30-90 minutes, irinotecan hydrochloride IV over 30 minutes, leucovorin calcium IV over 2 hours, and fluorouracil IV bolus followed by infusion over 46 hours on day 1. Treatment repeats every 2 weeks for at least 6 months in the absence of disease progression or unacceptable toxicity.
  * Group 3 (high topo-1 and both K-ras and BRAF wildtype): Patients are randomized to 1 of 3 treatment arms.

    * Arm I (regimen A [IrMdG]): Patients receive irinotecan hydrochloride, leucovorin calcium, and fluorouracil as in group 1, arm I.
    * Arm II (regimen C [IrOxMdG]): Patients receive irinotecan hydrochloride IV over 30 minutes, leucovorin calcium IV over 2 hours, oxaliplatin IV over 2 hours, and fluorouracil IV bolus followed by infusion over 46 hours on day 1. Treatment repeats every 2 weeks for at least 6 months in the absence of disease progression or unacceptable toxicity.
    * Arm III (regimen D [IrMdG and cetuximab]): Patients receive cetuximab, irinotecan hydrochloride, leucovorin calcium, and fluorouracil IV as in group 1, arm III.
  * Group 4 (high topo-1 and either K-ras or BRAF mutation): Patients are randomized to 1 of 3 treatment arms.

    * Arm I (regimen A [IrMdG]): Patients receive irinotecan hydrochloride, leucovorin calcium, and fluorouracil as in group 1, arm I.
    * Arm II (regimen C [IrOxMdG]): Patients receive irinotecan hydrochloride, leucovorin calcium, oxaliplatin, and fluorouracil as in group 3, arm II.
    * Arm III (regimen E [IrMdG and bevacizumab]): Patients receive bevacizumab, irinotecan hydrochloride, leucovorin calcium, and fluorouracil IV as group 2, arm III.

After completion of study therapy, patients are followed up periodically.

PROJECTED ACCRUAL: A total of 240 patients will be accrued for the feasibility study and approximately 3,000 patients will be accrued for the definitive study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal adenocarcinoma meeting 1 of the following criteria:

  * Prior or recurrent primary adenocarcinoma of the colon or rectum with clinical or radiological evidence of locally advanced or metastatic disease
  * Metastatic adenocarcinoma with clinical and/or radiological evidence of colorectal primary tumor
* Inoperable metastatic or locoregional disease

  * Patients suitable for surgical resection of metastatic disease after response to first-line or adjuvant chemotherapy not allowed and should be considered for the New-EPOC trial study
* Unidimensionally measurable disease (according to RECIST criteria)
* Must have completed adjuvant chemotherapy with fluorouracil +/- leucovorin calcium (FU +/- LC), capecitabine, or oxaliplatin combinations in the past 6 months

  * QUASAR 2 patients who have continued bevacizumab for 6 months following completion of chemotherapy are allowed immediately after completion of bevacizumab
* Rectal chemotherapy with FU +/- LC or capecitabine for allowed if completed ≥ 1 month ago
* Single tumor block available
* No brain metastasis

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Alkaline phosphatase ≤ 5 times upper limit of normal (ULN)
* Serum bilirubin ≤ 1.25 times ULN
* AST or ALT ≤ 2.5 times ULN
* Creatinine clearance ≥ 30 mL/min OR GFR ≥ 30 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Considered fit to undergo combination chemotherapy, with none of the following conditions:

  * Severe uncontrolled concurrent medical illness likely to interfere with protocol treatments, including any of the following:

    * Poorly controlled angina
    * Uncontrolled hypertension
    * Myocardial infarction within the past 3 months
  * History of severe peptic ulcer disease
  * Any psychiatric or neurological condition that is likely to compromise the patient's ability to give informed consent or to comply with oral medication
  * Nephrotic syndrome
  * Known coagulopathy
* No prior or current malignant disease that, in the judgement of the treating investigator, is likely to interfere with FOCUS 3 treatment or assessment of response
* No known hypersensitivity reactions to any of the components of the study treatments
* No personal or family history suggestive of dihydropyrimidine dehydrogenase (DPD) deficiency or with known DPD deficiency
* No history of uncontrolled seizures, central nervous system disorders, or psychiatric disability judged by the investigator to be clinically significant precluding informed consent
* Not able to attend or comply with treatment or follow-up scheduling

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior surgery
* No prior systemic chemotherapy for metastatic disease
* No ongoing therapy with cyclosporin-A
* No ongoing treatment with a contraindicated concomitant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3240 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Topoisomerase-1 (topo-1) and K-ras, BRAF results obtained within 10 working days after registration
Number of patients in which the interval between registration and randomization (RZ) is ≤ 10 days
Efficacy of fluorouracil with vs without irinotecan hydrochloride, fluorouracil, and leucovorin calcium (IrMdG) in low topo-1 tumors
Progression-free survival of patients with high topo-1 tumors treated with IrMdG with or without oxaliplatin
Efficacy of IrMdG with vs without cetuximab in K-ras wildtype tumors
Efficacy of IrMdG with vs without bevacizumab in K-ras mutant tumors

SECONDARY OUTCOMES:
Time from release of tumor block to receipt by pathology lab
If applicable, reason that RZ did not occur
Time from registration to treatment start
Time from data presentation to investigator to date of RZ
Reproducibility of K-ras, BRAF, and topo-1 results
Distribution frequencies
Costs of molecular testing
Toxicity according to NCI CTCAE v.3
Response rates
Progression-free survival
Attitudes of patients about tests and treatment

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Maughan, MD, Principal Investigator — Velindre NHS Trust
Locations (3):
- United Kingdom (3):
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Belfast City Hospital Trust Incorporating Belvoir Park Hospital, Belfast, Northern Ireland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales

REFERENCES:
- [Result] Maughan T, Wilson RH, Williams GT, et al.: Developing a biomarker-stratified trial design in advanced colorectal cancer: The MRC FOCUS 3 feasibility study. [Abstract] J Clin Oncol 29 (Suppl 15): A-TPS165, 2011.